CLINICAL TRIAL: NCT07402005
Title: Correlation of Lewis Erythrocyte Antigens With the Risk of Venous Thromboembolic Disease-VTE
Brief Title: The Correlation of Lewis Antigens With VTE
Status: Not yet recruiting | Type: Observational
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Eleftheria Lefkou, Assistant Professor of Transfusion Medicine, Larissa University Hospital
Other Study IDs: 52424
Record Dates: First submitted 2026-02-03; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Thromboembolic Disease
Keywords: VTE, LEWIS ANTIGEN
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with personal history of VTE: BLODD SAMPLING
- CONTROL GROUP- VOLUNTEERS BLOOD DONORS: CONTROL GROUP- HEALTHY BLOOD DONORS

SUMMARY:
The goal of this observational study is to learn if certain factors in a person's blood are linked to a history of venous thromboembolic disease (VTED), which includes conditions like deep vein thrombosis.

Lewis system antigens are natural markers found on red blood cells. Past research suggests that people without these specific markers might have a higher chance of developing heart disease, but the link to blood clots in veins is not well understood.

This study aims to answer:

* Are certain Lewis antigen types more common in people with a history of VTE?
* Do the Lewis antigen results relate to other known blood clot risk factors? Researchers will identify Lewis a and b antigens in 100 participants who attend the Haemostasis Disorders Clinic at the University Hospital of Larissa. All participants are people with a personal history of deep vein thrombosis, with or without an inherited or acquired tendency for blood clots.

Researchers will also record other known risk factors for VTED for each participant. This study is self-funded.

DETAILED DESCRIPTION:
Background Since 1992, research has reported a correlation between Lewis antigens and cardiovascular disease, primarily linked to increased endothelial activation in individuals who are Lewis a(-) b(-). Experimental studies in mice suggest an association between the FUT4 and FUT7 genes and the occurrence of venous thromboembolic disease (VTED), but there is a lack of in vivo studies on this subject in humans . This study aims to fill this knowledge gap by investigating this relationship in a clinical setting.

Study Objectives The primary objective is to investigate the relationship between Lewis system antigens and a personal history of VTED. The study will also assess the association between specific Lewis antigen phenotypes and other known risk factors for VTED.

Study Design This is an independent and self-funded, single-center, observational study (p. 1). Lewis a and b antigens will be identified serologically in a specific patient population, and these results will be correlated with existing clinical data on thrombophilia and other VTE risk factors Study Population and Setting The study will include 100 participants (goal sample size for 90% statistical power) with a personal history of deep vein thrombosis, regardless of whether they have hereditary or acquired thrombophilia . All participants are monitored at the Haemostasis Disorders Clinic of the Blood Transfusion Service at the University Hospital of Larissa, Greece. Written informed consent is obtained from all participants after they are fully informed about the study.

Methods and Outcome Measures Lewis antigens are identified using commercial reagents and gel cards from Grifols.

Primary Outcome Measure: The prevalence of different Lewis erythrocyte antigen phenotypes in patients with a history of VTED. (Time Frame: At the time of a single blood draw) Secondary Outcome Measure: The correlation between Lewis phenotypes and the presence of other known VTE risk factors or a confirmed diagnosis of thrombophilia. (Time Frame: Assessed using existing medical records at the time of a single blood draw) Statistical Analysis Statistical analysis will be performed using the SPSS software package.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-78 years with a personal history of deep venous thrombosis and/or Pulmonary Embolism.

Exclusion Criteria:1. Current pregnancy or postpartum period 2. Hepatic insufficiency 3. Alcoholic cirrhosis

-

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pateints with personal history of VTE
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to investigate the relationship between Lewis system antigens and venous thromboembolic disease (VTED). | From enrollment to the day of blood phenotyping- approximately 48 hours
  Lewis a and b antigens will be identified in patients with a personal history of deep vein thrombosis, with or without hereditary or acquired thrombophilia, who are being monitored at the Haemostasis Disorders Clinic of the Blood Transfusion Service of the University Hospital of Larissa. All patients, after being informed, will submit written consent for their participation in the study.
  Lewis antigens will be identified serologically using reagents and gel cards from Grifols. The results of the thrombophilia test and other known risk factors for VTE will be recorded. Statistical analysis will be performed using the SPSS package.
PRESENCE OF LEWIS A AND B ANTIGEN ON ERYTHROCYTE | From enrollment to the day of blood antigen phenotyping- approximately 48 hours
  NEGATIVE OR POSITIVE FOR LEWIS ANTIGENS

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Kotsi, MD, PhD, Study Chair — Blood Transfusion and Haemostasis Unit, Faculty Of Medicine, School Of Health Sciences, University of Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No
Our study does not plan to share Individual Participant Data (IPD) primarily due to strict limitations in the original informed consent process; participants did not grant permission for their data to be shared externally.

REFERENCES:
- [Background] Wang H, Morales-Levy M, Rose J, Mackey LC, Bodary P, Eitzman D, Homeister JW. alpha(1,3)-Fucosyltransferases FUT4 and FUT7 control murine susceptibility to thrombosis. Am J Pathol. 2013 Jun;182(6):2082-93. doi: 10.1016/j.ajpath.2013.02.010. Epub 2013 Apr 2. PMID 23562273
- [Background] Hein HO, Sorensen H, Suadicani P, Gyntelberg F. The Lewis blood group--a new genetic marker of ischaemic heart disease. J Intern Med. 1992 Dec;232(6):481-7. doi: 10.1111/j.1365-2796.1992.tb00620.x. PMID 1474347
- [Background] Ellison RC, Zhang Y, Myers RH, Swanson JL, Higgins M, Eckfeldt J. Lewis blood group phenotype as an independent risk factor for coronary heart disease (the NHLBI Family Heart Study). Am J Cardiol. 1999 Feb 1;83(3):345-8. doi: 10.1016/s0002-9149(98)00866-2. PMID 10072221
- [Background] Salomaa V, Pankow J, Heiss G, Cakir B, Eckfeldt JH, Ellison RC, Myers RH, Hiller KM, Brantley KR, Morris TL, Weston BW. Genetic background of Lewis negative blood group phenotype and its association with atherosclerotic disease in the NHLBI family heart study. J Intern Med. 2000 Jun;247(6):689-98. doi: 10.1046/j.1365-2796.2000.00682.x. PMID 10886491
- [Background] Bharath R, Nair KKM, Gupta D, Vijayan R. Assessment of Lewis negative phenotype as a risk factor for multivessel disease in patients with acute coronary syndrome. Transfus Clin Biol. 2022 May;29(2):129-133. doi: 10.1016/j.tracli.2021.12.008. Epub 2021 Dec 30. PMID 34974187
- See also: University Hospital of Larissa, Thessaly — https://www.uhl.gr/
- Available data/document: Study Protocol: 52424 — https://www.uhl.gr/ — https://www.uhl.gr/

DOCUMENTS (1):
  • Informed Consent Form (2026-01-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT07402005/ICF_000.pdf